CLINICAL TRIAL: NCT06554314
Title: Effect of Probiotics on Regulating Gut Health and Blood Lipid in Overweight and Obese Adults
Brief Title: Effect of Probiotics on Regulating Gut Health and Blood Lipid in Adults
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chung Shan Medical University (Other)
Collaborators: Nutrarex Biotech Ltd. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: CS2-23191
Record Dates: First submitted 2024-08-12; First posted 2024-08-15 (Actual); Last update posted 2024-08-15 (Actual); Status verified 2024-08

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity | interventions — Probiotics

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Probiotics (Experimental): Probiotic capsules, 300 mg each, one daily for a total of 300 mg for 4 weeks
  Interventions: Dietary Supplement: probiotics
- Placebo (Placebo Comparator): The placebo capsules had the same composition as the experimental capsules, except that they did not contain probiotics, and should be used for 4 weeks.
  Interventions: Dietary Supplement: probiotics

INTERVENTIONS:
Dietary Supplement: probiotics — Eat a capsule for once, and once a day

SUMMARY:
The purpose of this study was to evaluate the efficacy of 1 capsules (300 mg per capsule) of Nutrarex Probiotic Capsules per day in regulating gut health and blood lipid in adults by clinical trial.

DETAILED DESCRIPTION:
This experiment is carried out in a controlled manner. Before the subjects enter the research experiment, they need to follow their original lifestyle. The habits of maintaining a constant body weight for more than 2 weeks before the test, such as calorie balance in the diet and the amount of activity. Then enter the test to carry out the evaluation test of probiotics to the end. 50 subjects were randomized, 25 to placebo and 25 to probiotics. The subjects took one capsules of Nutrarex probiotics daily, a total of 300 mg. Continue to take it for 4 weeks, and perform blood routine tests. Body composition detection, waist and hip circumference measurement, related index analysis and 24-hour dietary questionnaires, gut health questionnaires and stool samples were collected and analyzed for 4 weeks before and after treatment.

ELIGIBILITY:
Inclusion Criteria:

* male or female participants
* aged 20-65 years old
* body mass index in 25-27 kg/m2 or body fat > 25% for men and > 30% for women

Exclusion Criteria:

* cancer, chronic heart disease, use drugs which pharmacological effects may affect immunity having systemic infections
* using probiotics.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-05-17 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-05-31 (Estimated)

PRIMARY OUTCOMES:
Change from baseline serum lipids at week 4 | Week0, Week4
  Compared the difference of serum lipids level between the week 4 and 0

CONTACTS AND LOCATIONS:
Overall Officials: Yin-Chin Liu, MS student, Principal Investigator — Chung Shan Medical University
Locations (1):
- Chung Shan Medical University, Taichung, South, Taiwan